CLINICAL TRIAL: NCT06534996
Title: A Single Arm Pilot Study of the Chinese Herbal Medicine Formula (SCD-2101) for the Functional Constipation in the Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Professor, Hong Kong Baptist University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/23-24/0482
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Functional Constipation
Keywords: elderly, Chinese Herbal Medicine, Functional Constipation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): During the 2-week intervention, all participants are required to take 150ml of SCD-2101 liquid (a Chinese herbal medicine formula containing four herbs) twice per day
  Interventions: Drug: SCD-2101

INTERVENTIONS:
Drug: SCD-2101 — Tradictional Chinese Medicine formula (SCD-2101)

SUMMARY:
This single-arm, open-label pilot clinical trial will test the hypothesis that SCD-2101, a Chinese herbal medicine formula, will have efficacy in alleviating constipation in elderly individuals with functional constipation. All participants (n=14) will receive 2 weeks of intervention and 2 weeks of follow-up.

DETAILED DESCRIPTION:
Purpose of the Study: This clinical study aims to observe the efficacy and safety of treating functional constipation in the elderly with the traditional Chinese medicine formula SCD-2101.

Study Design: Single-arm, pilot clinical trial.

Target Population: Patients aged 60 years or above, meeting the Rome IV diagnostic criteria for functional constipation, with no more than 2 Complete Spontaneous Bowel Movements (CSBM) per week, capable of understanding and using Chinese, and have signed the informed consent form.

Sample Size: This clinical trial is an exploratory study, with an estimated sample size of 14 participants.

Treatment Plan: Participants will take the traditional Chinese medicine compound decoction for two weeks, twice a day, 150 milliliters each time, after meals.

Primary Outcome: Response rate of Complete Spontaneous Bowel Movements (CSBM) (Time point: end of 2-week treatment)

Secondary Outcomes:

1. Change in the number of Complete Spontaneous Bowel Movements (CSBM) per week compared to baseline (Time point: end of 2-week treatment)
2. Change in the number of Spontaneous Bowel Movements (SBM) per week compared to baseline (Time point: end of 2-week treatment)
3. Types and severity of adverse reactions after taking the medication

Safety Outcomes:

1. Any adverse reaction symptoms/adverse events occurring after the trial treatment
2. General physical examination items (including heart rate, blood pressure, etc.)

Statistical Analysis: The database is constructed using REDCap, and all statistics are analyzed using SPSS version 23 statistical analysis software, to analyze the general conditions, demographic and other baseline characteristics, compliance, efficacy, and safety of the participants.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 60 years old (2) Meet the Rome IV diagnostic criteria for functional constipation (3) Complete spontaneous bowel movements ≤ 2 times per week, to be assessed based on a 2-week electronic diary record (CSBMs are defined as the number of times within a 24-hour period that the patient can defecate spontaneously without the use of laxatives or enemas and feels that the stool is completely evacuated) (4) Have colonoscopy results with a diagnosis of no significant abnormalities seen or no more than 3 colorectal polyps, each less than 0.5 cm in size (based on results within the last 5 years before screening) (5) Understand and be able to follow written and oral instructions in Chinese (6) Capable of independently using WhatsApp and an electronic diary, and completing a 2-week electronic diary record during the screening period (7) The subject is informed and voluntarily signs the informed consent form.

Exclusion Criteria:

* (1) Secondary constipation (constipation caused by drugs or other diseases); (2) Currently using or requiring continued use of medications that may affect the outcomes of the trial (including but not limited to: antibiotics, hormonal drugs, analgesics, neurotransmitter drugs, gut flora-regulating medications, etc.); (3) Colonoscopy or sigmoidoscopy reveals clinically significant abnormalities; (4) Clinically significant abnormalities in laboratory tests or imaging examinations within the last 6 months; (5) History of allergy to traditional Chinese medicine; (6) History of abdominal surgery within the past year (except for laparoscopic appendectomy); (7) Patients with psychiatric diseases or those requiring the use of psychotropic drugs; (8) Deemed by the researchers as unsuitable to participate in this study for psychological or physical reasons.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Response rate of Complete Spontaneous Bowel Movements (CSBM) | from baseline to Week 2
  A CSBM responder is defined as a patient who meets the CSBM responder criterion (i.e., a mean increase of CSBM≥1/week compared with CSBM at baseline, in at least 2 out of 4 weeks). A spontaneous bowel movement (SBM) is defined as a bowel movement without laxative use in the preceding 24 hours. A CSBM is defined as a SBM that is associated with a sense of complete evacuation. Baseline of weekly CSBM will be the average between Week -2 and Week 0.

SECONDARY OUTCOMES:
Change in the number of Complete Spontaneous Bowel Movements (CSBM) per week compared to baseline | from baseline to Week 2
  A spontaneous bowel movement (SBM) is defined as a bowel movement without laxative use in the preceding 24 hours. A CSBM is defined as a SBM that is associated with a sense of complete evacuation. Baseline of weekly CSBM will be the average between Week -2 and Week 0.
Change in the number of Spontaneous Bowel Movements (SBM) per week compared to baseline | from baseline to Week 2
  weekly Spontaneous Bowel Movement (SBM)
Types and severity of adverse reactions after taking the medication | from baseline to Week 2
  Assessed by number of adverse events or side effects

OTHER OUTCOMES:
Safety Outcomes: (1) Any adverse reaction symptoms/adverse events occurring after the trial treatment | from baseline to Week 2
  Assessed by number of adverse events or side effects
Safety Outcomes: (2) General physical examination items (including heart rate, blood pressure, etc.) | from baseline to Week 2
  Assessed by number of adverse events or side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Baptist University, Kowloon Tong, Hong Kong